CLINICAL TRIAL: NCT01471652
Title: Chronic Fatigue Syndrome: Correction of Mitochondrial Dysfunction by Conditioning Exercise and Nutraceutical Therapy.
Brief Title: Chronic Fatigue Syndrome: A Presumptive Mitochondrial Disorder
Acronym: CFS:M
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAJ0702
Record Dates: First submitted 2011-11-09; First posted 2011-11-15 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Fatigue Syndrome
Keywords: myalgic encephalopathy; chronic fatigue syndrome; post viral infection; fatigue; muscle pain; unrefreshing sleep; fuzzy thought; poor memory; forgetfulness
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Myalgia; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutraceuticals (Active Comparator): Subjects will receive a combination of 4 nutraceuticals (CoEnzyme Q10, acetyl-L-carnitine, alpha-lipoic acid, docosahexaenoic acid (DHA)) and a multivitamin.
  Interventions: Drug: Nutraceutical supplements
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nutraceutical supplements — 1. CoEnzyme Q10: oral gel capsule bid
  2. Acetyl L-carnitine: oral capsule bid
  3. Alpha Lipoic Acid: oral tablet qd
  4. Docosahexaenoic acid: oral gel capsule bid
  Arms: Nutraceuticals
Drug: Placebo — Capsule form to imitate the following nutraceuticals:
  1. Placebo 1: oral gel capsule bid
  2. Placebo 2: oral capsule bid
  3. Placebo 3: oral tablet qd
  4. Placebo 4: oral gel capsule bid
  Arms: Placebo

SUMMARY:
The pathogenesis of chronic fatigue syndrome (CFS) is poorly understood and no effective therapy has been developed. Recent studies suggest that a preceding viral infection causes mitochondrial dysfunction of the brain and skeletal muscle of genetically susceptible individuals. There is no specific laboratory test to identify patients with CFS. However, certain clinical manifestations are similar to those seen in mitochondrial disorders. Both patients with mitochondrial disorders and CFS manifest elevated serum lactate levels after exercise, and demonstrate elevated brain cerebrospinal fluid levels and decreased brain glutathione levels on nuclear magnetic resonance (NMR) spectroscopy.

Therapy consisting of daily conditioning exercise, dietary recommendations, and nutraceutical supplements (ENT) has been show to be beneficial in treating patients with mitochondrial disorders. Similar therapy has been instituted in individual patients with CFS and has been shown to also improve their clinical conditions.

A placebo-controlled trial will be undertaken in 24 CFS patients aged 25-55. Patients fulfilling the CDC criteria for CFS will participate in this 6 month study. Other medical causes for fatigue will be excluded. Half the patients will receive treatment consisting of daily conditioning exercise plus nutraceutical supplements (ENT), that has been shown to be beneficial for patients with mitochondrial dysfunction, while the other half will receive daily conditioning exercise and placebo tablets. Response to ENT will be evaluated by maximum oxygen consumption (VO2max) and circulating lactate levels during & after treadmill exercise, a 6-minute walk test, and a fatigue questionnaire. In addition, whether ENT corrects the elevated brain cerebrospinal fluid levels and decreased brain glutathione levels will be measured. To ensure compliance to therapy patients will be monitored frequently. The objective of this study is to assess the safety and efficacy of ENT and whether ENT leads to sustained improvement of CFS patients compared to their baseline status, and compared to an exercised group of patients not receiving supplements.

DETAILED DESCRIPTION:
Chronic fatigue syndrome (CFS), also known as myalgic encephalitis (ME), is clinically characterized as a multisystem illness exhibiting debilitating fatigue, musculoskeletal pain, disturbed sleep, and impaired memory and concentration. Its diagnosis is non-specific and symptom based, with no real biomarkers yet identified. The etiology and pathophysiology of CFS remain obscure. There is a long-standing hypothesis that individuals with CFS have normal metabolism and their fatigue is psychological, with energy being wasted through the processes of anxiety, stress, and depression. The more CFS is investigated, however, the clearer it becomes that this is incorrect, and that it is probably a metabolic dysfunction resulting in insufficient energy production. A number of studies have suggested that there may be a genetic contribution to CFS. In addition, a severe viral illness frequently predisposes the onset of CFS, while a number of pathogens have been linked to CFS (2, 3, 6). Although some patients develop CFS after an acute infection such as mononucleosis, some investigators believe it arises from the reactivation of a latent virus in the host, both resulting in a chronic low-level activation of the immune system.

As more data are acquired, we and others believe that CFS is actually a metabolic mitochondrial dysfunction resulting in insufficient energy production. Mounting evidence indicates that viral infections in genetically susceptible individuals can cause changes in mitochondrial function. Many features observed in CFS are similar to those seen in genetic mitochondrial disorders. Firstly, some muscle biopsies in patients with CFS have shown both abnormal mitochondrial degeneration and severe deletions of mitochondrial DNA genes. Mitochondrial dysfunction increases the production of free radicals and reactive oxygen species (ROS), which cause oxidative damage, believed to contribute to CFS pathogenesis. Carnitine is required for metabolic reactions including mitochondrial fatty acid oxidation. A deficiency of serum acylcarnitine has been observed in CFS patients, suggesting that there is increased utilization of carnitine in CFS, thereby decreasing energy production. In mitochondrial disorders, utilization of pyruvate is decreased, resulting in higher circulating and muscle levels of lactate, as well as decreased oxidative phosphorylation and energy production. Brain ventricular cerebrospinal lactate is elevated, and brain glutathione is decreased, in both mitochondrial disorders and CFS. In CFS patients cerebrospinal lactate is increased by approximately 300% compared to that found in generalized anxiety disorder and healthy individuals. Using brain NMR spectroscopy, the distinction between CFS and psychological disorders can be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the criteria for CFS of the US Centers for Disease Control and Prevention (CDC), which requires persistent, unexplained fatigue for at least 6 months, concurrent with four of the following:

* impaired memory/concentration
* sore throat, new headaches
* unrefreshing sleep, muscle pain
* multi-joint pain
* tender lymph nodes
* post-exertional malaise

As well, due to the frequency of visits subjects must currently reside in the greater New York area.

Exclusion Criteria:

* shortness of breath
* heart disease
* high blood pressure
* other severe chronic illnesses
* clinical depression
* generalized anxiety disorder
* insomnia
* inflammatory arthritis
* anemia
* hypothyroidism
* other conditions associated with significant fatigue
* history of alcohol, tobacco, or drug abuse

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in rate of fatigue status and other CFS symptoms | 0, 3, and 6 months
  Rate of decrease in fatigue and other CFS symptoms, as measured by SF-36 and The Fatigue Assessment Instrument.

SECONDARY OUTCOMES:
Change in brain lactate and glutathione levels | 0 and 6 months
  Patients will undergo nuclear magnetic resonance spectroscopy of the brain prior to starting therapy (baseline) and repeat it after 6 months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred E Slonim, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Department of Clinical Genetics, New York, New York, United States